CLINICAL TRIAL: NCT04813263
Title: A Post-marketing Observational Study for Venetoclax in Patients Diagnosed With Acute Myeloid Leukemia in Japan
Brief Title: Study of Oral Venetoclax Tablets to Evaluate Adverse Events and Change in Disease Activity in Participants of Any Age With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-408
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute Myeloid Leukemia (AML); Cancer; Venetoclax; Venclexta; Venclyxto
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Treated With Venetoclax: Participants who are administrated venetoclax for treatment of AML under routine clinical practice.

SUMMARY:
Acute Myeloid Leukemia (AML) is an aggressive and rare cancer of myeloid cells (a white blood cell responsible for fighting infections) and is the most common acute leukemia in adults. This study will assess how safe and effective oral venetoclax is in participants with AML. Adverse events and change in disease activity will be monitored under routine clinical practice.

Venetoclax is an approved drug to treat Acute Myeloid Leukemia (AML). Around 400 participants of any age who are treated with oral venetoclax tablets for AML in accordance with the approved label will be enrolled in the study across Japan.

Participants will be followed up to 52 weeks following the first dose of oral venetoclax tablets.

There is expected to be no additional burden for participants in this study. Data will be collected by information provided by participating physicians based on routine medical records.

ELIGIBILITY:
Inclusion Criteria:

- All participants who are administered venetoclax for treatment of AML.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who are prescribed venetoclax for the treatment of Acute Myeloid Leukemia (AML) in routine clinical practice across Japan.
Sampling Method: Non-Probability Sample
Enrollment: 424 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With ≥ Grade 3 Neutropenia of Venetoclax Regimens With Unfit Acute Myeloid Leukemia (AML) | Up to 52 weeks.
  Percentage of participants with a high grade (≥ Grade 3) protocol specified neutropenia during and after treatment with venetoclax.

SECONDARY OUTCOMES:
Percentage of Participants With Febrile Neutropenia and Thrombocytopenia | Up to 52 weeks
  Percentage of participants with protocol specified febrile neutropenia and thrombocytopenia during and after treatment with venetoclax.
Percentage of Participants With Tumor Lysis Syndrome (TLS) | Up to 52 weeks
  Percentage of participants with protocol specified TLS during and after treatment with venetoclax.
Percentage of Participants Reported >= Grade 3 Adverse Events (AE)/Adverse Drug Reactions (ADR) | Up to 52 weeks
  Grade 3 and above AE/ADR are serious adverse event (SAE) that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above.
Percentage of Participants Reported Adverse Events (AE)/Adverse Drug Reaction (ADR) | Up to 52 weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either definitely related, probably related, possibly related or unrelated.
Percentage of Participants With AE/ADR When Used Concomitantly With CYP3A Inhibitors or Growth Colony Stimulating Factor (G-CSF) | Up to 52 weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either definitely related, probably related, possibly related or unrelated.
Percentage of Participants With Composite Complete Remission Rate (CR + CRi) | Up to 52 weeks
  Composite Complete remission (CRc) is defined as Complete Remission (CR) + CRi (CR with incomplete blood count recovery) based on protocol criteria.
Median Time to Best Response | Up to 52 weeks.
  Time to Best Response is measured as the time in months from the first dose of study treatment to the date of first documented documentation of a confirmed response of partial response (PR) or better.
Median Treatment Duration | Up to 52 weeks
  Median time for duration of oral venetoclax treatment in participants with Acute Myeloid Leukemia.
Median Overall Survival | Up to 52 weeks
  Time from the date of first oral Venetoclax intake to the date of death from any cause.
Median Duration of Composite Complete Remission | Up to 52 weeks
  Time from the date of first oral Venetoclax intake and the date of the assessment having documented Complete Remission with incomplete Hematologic recovery (CRi).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (281):
- Japan (281):
  - Anjou Kousei Hospital /ID# 244213, Anjo-shi, Aichi-ken
  - Nagoya City West Medical Center /ID# 250844, Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital /ID# 243785, Nagoya, Aichi-ken
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital /ID# 242173, Nagoya, Aichi-ken
  - Nagoya University Hospital /ID# 246009, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 256177, Nagoya, Aichi-ken
  - National Center for Geriatrics and Gerontology /ID# 251683, Obu-shi, Aichi-ken
  - Toyohashi Municipal Hospital /ID# 243784, Toyohashi, Aichi-ken
  - Toyokawa City Hospital /ID# 242707, Toyokawa-shi, Aichi-ken
  - Toyota Memorial Hospital /ID# 242175, Toyota-shi, Aichi-ken
  - Akita city Hospital /ID# 240008, Akita, Akita
  - Odate Municipal General Hospital /ID# 258238, Odate-shi, Akita
  - Aomori Prefectural Central Hospital /ID# 249442, Aomori, Aomori
  - National Hospital Organization Hirosaki General Medical Center /ID# 246008, Hirosaki-shi, Aomori
  - Asahi General Hospital /ID# 233889, Asahi-shi, Chiba
  - Chiba Aoba Municipal Hospital /ID# 240565, Chiba, Chiba
  - Chiba University Hospital /ID# 246011, Chiba, Chiba
  - Duplicate_Chiba Cancer Center /ID# 248122, Chiba, Chiba
  - KK Clinic Ichihara /ID# 250859, Ichihara, Chiba
  - Chiba Rosai Hospital /ID# 238767, Ichihara-shi, Chiba
  - Tokyo Dental College Ichikawa General Hospital /ID# 262626, Ichikawa-shi, Chiba
  - Nippon Medical Chiba Hokusoh Hospital /ID# 250297, Inzai-shi, Chiba
  - Kameda General Hospital /ID# 241877, Kamogawa-shi, Chiba
  - The Jikei University Kashiwa Hospital /ID# 259510, Kashiwa-shi, Chiba
  - National Cancer Center Hospital East /ID# 241917, Kashiwa-shi, Chiba
  - Kimitsu Chuo Hospital /ID# 248776, Kisarazu-shi, Chiba
  - Chiba West General Hospital /ID# 262918, Matsudo-shi, Chiba
  - Tsudanuma Central General Hospital /ID# 245890, Narashino-shi, Chiba
  - Japanese Red Cross Narita Hospital /ID# 243775, Narita-shi, Chiba
  - IUHW Narita Hospital /ID# 240574, Narita-shi, Chiba
  - Chibaken Saiseikai Narashino Hospital /ID# 254491, Narshino-shi, Chiba
  - Toho University Sakura Medical Center /ID# 252187, Sakura-shi, Chiba
  - Watanabe Hospital /ID# 254476, Matsuyama, Ehime
  - Ehime Prefectural Central Hospital /ID# 261348, Matsuyama, Ehime
  - Matsuyama Shimin Hospital /ID# 243050, Matsuyama, Ehime
  - National Hospital Organization Shikoku Cancer Center /ID# 242171, Matsuyama, Ehime
  - Ehime University Hospital /ID# 244207, Toon-shi, Ehime
  - Fukuiken Saiseikai Hospital /ID# 245062, Fukui-shi, Fukui
  - Fukuiken Saiseikai Hospital /ID# 246005, Fukui-shi, Fukui
  - Saiseikai Fukuoka Genaral Hospital /ID# 255193, Fukuoka, Fukuoka
  - National Hospital Organization Kyushu Medical Center /ID# 242026, Fukuoka, Fukuoka
  - Fukuoka Wajiro Hospital /ID# 238755, Fukuoka, Fukuoka
  - National Hospital Organization Kyushu Cancer Center /ID# 244217, Fukuoka, Fukuoka
  - Kyushu University Hospital /ID# 248781, Fukuoka, Fukuoka
  - Fukuoka University Hospital /ID# 244214, Fukuoka, Fukuoka
  - Japanese Red Cross Fukuoka Hospital /ID# 241181, Fukuoka, Fukuoka
  - Murakami Karindoh Hospital /ID# 256179, Fukuoka, Fukuoka
  - Aso Iizuka Hospital /ID# 266806, Iizuka, Fukuoka
  - NHO Kokura Medical Center /ID# 257008, Kitakyusyu-shi, Fukuoka
  - Wakamatsu Hospital /ID# 251728, Kitakyusyu-shi, Fukuoka
  - Shinkoga Hospital /ID# 248786, Kurume, Fukuoka
  - Kurume University Hospital /ID# 240885, Kurume-shi, Fukuoka
  - St. Mary's Hospital /ID# 242332, Kurume-shi, Fukuoka
  - Omuta City Hospital /ID# 246823, Omuta-shi, Fukuoka
  - Nagata Hospital /ID# 256180, Yanagawa-shi, Fukuoka
  - Kita Fukushima Medical Center /ID# 250296, Date-shi, Fukushima
  - Fukushima Minami Cardiovascular Hospital /ID# 252216, Fukushima, Fukushima
  - Tokiwakai Jyoban Hospital /ID# 257007, Iwaki, Fukushima
  - Iwaki Kyoritsu General Hospital /ID# 260209, Iwaki, Fukushima
  - Ohta Nishinouchi Hospital /ID# 243052, Koriyama-shi, Fukushima
  - Shirakawa Kosei General Hosp. /ID# 245815, Shirakawa-shi, Fukushima
  - Gifu Municipal Hospital /ID# 241156, Gifu, Gifu
  - Gifu University Hospital /ID# 241183, Gifu, Gifu
  - Gifu Red Cross Hospital /ID# 240562, Gifu, Gifu
  - Ogaki Municipal Hospital /ID# 239353, Ogaki-shi, Gifu
  - Japanese Red Cross Takayama Hospital /ID# 240568, Takayama, Gifu
  - Fujioka General Hospital /ID# 255196, Fujioka-shi, Gunma
  - Gunmaken Saiseikai Maebashi Hospital /ID# 239383, Maebashi, Gunma
  - Gunma Prefectural Cancer Center /ID# 242177, Ota-shi, Gunma
  - National Hospital Organization Shibukawa Medical Center /ID# 245026, Shibukawa-shi, Gunma
  - Tatebayashi Kosei General Hospital /ID# 252188, Tatebayashi-shi, Gunma
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital /ID# 240880, Hiroshima, Hiroshima
  - Mihara Shiromachi Hospital /ID# 246754, Mihara, Hiroshima
  - NHO Hiroshima-Nishi Medical center /ID# 238766, Otake-shi, Hiroshima
  - Kitami Red Cross Hospital /ID# 251065, Kitami-shi, Hokkaido
  - Steel Memorial Muroran Hospita /ID# 231383, Muroran-shi, Hokkaido
  - Obihiro kosei Hospital /ID# 252218, Obihiro-shi, Hokkaido
  - Sapporo Hokuyu Hospital /ID# 250856, Sapporo, Hokkaido
  - Homecareclinicn-Consept /Id# 239377, Sapporo, Hokkaido
  - Hokkaido Cancer Center /ID# 249441, Sapporo, Hokkaido
  - Sapporo Hokushin Hospital /ID# 241878, Sapporo, Hokkaido
  - Sapporo Kiyota Hospital /ID# 231385, Sapporo, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 249446, Sapporo, Hokkaido
  - Sapporo Medical University Hospital /ID# 252217, Sapporo, Hokkaido
  - Hokkaido University Hospital /ID# 244223, Sapporo, Hokkaido
  - Aiiku Hospital /ID# 239047, Sapporo, Hokkaido
  - Tenshi Hospital /ID# 243051, Sapporo, Hokkaido
  - Sunagawa City Medical Center /ID# 239382, Sunagawa, Hokkaido
  - Wakkanai City Hospital /ID# 243782, Wakkanai, Hokkaido
  - Ako Central Hospital /ID# 239721, Ako-shi, Hyōgo
  - Hyogo Prefectural Amagasaki General Medical Center /ID# 239355, Amagasaki-shi, Hyōgo
  - Itami City Hospital /ID# 233888, Itami-shi, Hyōgo
  - Hyogo Prefectural Kobe Children's Hospital /ID# 245817, Kobe, Hyōgo
  - Kobe City Medical Center General Hospital /ID# 246010, Kobe, Hyōgo
  - Shinko Hospital /ID# 233782, Kobe, Hyōgo
  - Konan Medical Center /ID# 246079, Kobe, Hyōgo
  - Hyogo?Prefectural?Nishinomiya Hospital /ID# 239354, Nishinomiya-shi, Hyōgo
  - Hyogo Medical University Hospital /ID# 240569, Nishinomiya-shi, Hyōgo
  - Kita-harima Medical Center /ID# 254490, Ono-shi, Hyōgo
  - Hyogo Prefectural Tamba Medical Center /ID# 240884, Tamba-shi, Hyōgo
  - Hyogo College of Medicine Sasayama Medical Center /ID# 240888, Tanbasasayama-shi, Hyōgo
  - Hyogo Prefectural Awaji Medical Center /ID# 240823, 洲本市, Hyōgo
  - National Hospital Organization Mito Medical Center /ID# 239719, Higashi Ibaraki-gun, Ibaraki
  - Hitachi General Hospital /ID# 239376, Hitachi-shi, Ibaraki
  - JA Toride Medical Center /ID# 240573, Toride-shi, Ibaraki
  - University of Tsukuba Hospital /ID# 242023, Tsukuba, Ibaraki
  - JCHO Kanazawa Hospital /ID# 239379, Kanazawa, Ishikawa-ken
  - Iwate Prefectural Isawa Hospital /ID# 246819, Oshu-shi, Iwate
  - Iwate Medical University Hospital /ID# 251009, Shiwa-gun, Iwate
  - Sakaide City Hospital /ID# 240563, Sakaidechō, Kagawa-ken
  - Imakiire General Hospital /ID# 258237, Kagoshima, Kagoshima-ken
  - Imamura General Hospital /ID# 234006, Kagoshima, Kagoshima-ken
  - Medical Corporation Seijinkai Ikeda Hospital /ID# 242174, Kanoya-shi, Kagoshima-ken
  - Shonan Tobu Sogo Hospital /ID# 241913, CHIGASAKI-shi, Kanagawa
  - Shonan Kamakura General Hospital /ID# 243053, Kamakura-shi, Kanagawa
  - Teikyo University Mizonokuchi Hospital /ID# 244842, Kawasaki, Kanagawa
  - Kawasaki Municipal Hospital /ID# 241162, Kawasaki-shi, Kanagawa
  - Japan Organization of Occupational Health and Society Kanto Rosai Hospital /ID# 255195, Kawasaki-shi, Kanagawa
  - Toranomon Hospital Kajigaya /ID# 256186, Kawasaki-shi, Kanagawa
  - Yokohama City University Medical Center /ID# 248777, Yokohama, Kanagawa
  - Saiseikai Yokohamashi Nanbu Hospital /ID# 247955, Yokohama, Kanagawa
  - St. Marianna University School of Medicine Yokohama City Seibu Hospital /ID# 266803, Yokohama, Kanagawa
  - Kanagawa Cancer Center /ID# 246822, Yokohama, Kanagawa
  - Kochi Health Sciences Center /ID# 241182, Kochi, Kochi
  - National Hospital Organization Kumamoto Medical Center /ID# 240886, Kumamoto, Kumamoto
  - Kumamoto University Hospital /ID# 239720, Kumamoto, Kumamoto
  - Kumamoto Shinto General Hospital /ID# 242176, Kumamoto, Kumamoto
  - Kumamoto City Hospital /ID# 254494, Kumamoto-shi,Kumamoto, Kumamoto
  - Kumamoto Kenhoku Hospital /ID# 258240, Tamana-shi, Kumamoto
  - Kumamoto Minami National Hospital /ID# 242169, Uki, Kumamoto
  - JCHO Kumamoto General Hospital /ID# 248779, Yatsushiro, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine /ID# 244843, Kyoto, Kyoto
  - JCHO Kyoto Kuramaguchi Medical /ID# 248775, Kyoto, Kyoto
  - Japanese Red Cross Kyoto Daiichi Hosital /ID# 248124, Kyoto, Kyoto
  - Kyoto University Hospital /ID# 244844, Kyoto, Kyoto
  - National Hospital Organization Kyoto Medical Center /ID# 239092, Kyoto, Kyoto
  - Uji Tokushukai Medical Center /ID# 241876, Uji-shi, Kyoto
  - Takeuchi Hospital /ID# 238750, Tsu, Mie-ken
  - Miyagi Cancer Center /ID# 241879, Natori-shi, Miyagi
  - Osaki Citizen Hospital /ID# 249447, Osaki-shi, Miyagi
  - Miyagi Chuo Hospital /ID# 259511, Sendai, Miyagi
  - Tohoku University Hospital /ID# 243757, Sendai, Miyagi
  - National Hospital Organization Sendai Medical Center /ID# 239384, Sendai, Miyagi
  - Miyazaki Prefectural Miyazaki Hospital /ID# 251730, Miyazaki, Miyazaki
  - Koga General Hospital /ID# 248120, Miyazaki, Miyazaki
  - University of Miyazaki Hospital /ID# 248805, Miyazaki, Miyazaki
  - Miyazaki Prefectural Nobeoka Hospital /ID# 248715, Nabeoka-shi, Miyazaki
  - Nagasaki Goto Chuoh Hospital /ID# 239723, Goto-shi, Nagasaki
  - Jap Red Cross Nagasaki Genbaku /ID# 245029, Nagasaki, Nagasaki
  - Nagasaki University Hospital /ID# 245028, Nagasaki, Nagasaki
  - NHO Nagasaki Medical Center /ID# 240571, Omura-shi, Nagasaki
  - Sasebo City General Hospital /ID# 238759, Sasebo-shi, Nagasaki
  - Nara Hospital Kinki University Faculty of Medicine, /ID# 250295, Ikoma-shi, Nara
  - Nara Medical University Hospital /ID# 251726, Kashihara-shi, Nara
  - Nara Prefecture General Medical Center /ID# 254492, Nara, Nara
  - Tenri Hospital /ID# 250855, Tenri-shi, Nara
  - Niigata University Medical & Dental Hospital /ID# 245027, Niigata, Niigata
  - National Hospital Organization Beppu Medical Center /ID# 247894, Beppu-shi, Oita Prefecture
  - Kyushu University Beppu Hospital /ID# 249444, Beppu-shi, Oita Prefecture
  - Oita Memorial Hospital /ID# 246818, Ōita, Oita Prefecture
  - Oita Prefectural Hospital /ID# 243786, Ōita, Oita Prefecture
  - Almeida Memorial Hospital /ID# 241916, Ōita, Oita Prefecture
  - Oita University Hospital /ID# 261976, Yufu, Oita Prefecture
  - Kawasaki Medical School Hospital /ID# 242709, Kurashiki-shi, Okayama-ken
  - Kurashiki Central Hospital /ID# 244205, Kurashiki-shi, Okayama-ken
  - Kaneda Hospital /ID# 238757, Maniwa, Okayama-ken
  - Duplicate_Okayama University Hospital /ID# 240887, Okayama, Okayama-ken
  - Duplicate_Okayama University Hospital /ID# 243755, Okayama, Okayama-ken
  - Japanese Red Cross Okayama Hospital /ID# 240879, Okayama, Okayama-ken
  - Okayama Medical Center /ID# 243759, Okayama, Okayama-ken
  - Naha City Hospital /ID# 242027, Naha, Okinawa
  - University of the Ryukyus Hospital /ID# 246821, Nakagami-gun, Okinawa
  - Nakagami Hospital /ID# 243787, Okinawa-shi, Okinawa
  - Shiroyama Hospital /ID# 246762, Habikino-shi, Osaka
  - Ishikiriseiki Hospital /ID# 246077, Higashiosaka, Osaka
  - Kansai Medical University Hospital /ID# 246820, Hirakata-shi, Osaka
  - Izumi City General Hospital /ID# 253204, Izumi-shi, Osaka
  - Osaka Women's and Children's Hospital /ID# 266805, Izumi-Shi, Osaka
  - Kishiwada City Hospital /ID# 234002, Kishiwada-shi, Osaka
  - Sumitomo Hospital /ID# 243774, Kita-ku, Osaka
  - Seijukai Hospital /ID# 248788, Neyagawa, Osaka
  - Osaka Saiseikai Nakatsu Hospital /ID# 244209, Osaka, Osaka
  - Kitano Hospital /ID# 248785, Osaka, Osaka
  - Osaka City General Hospital /ID# 244210, Osaka, Osaka
  - National Hospital Organization Osaka National Hospital /ID# 238764, Osaka, Osaka
  - Otemae Hospital /ID# 250857, Osaka, Osaka
  - Osaka International Cancer Institute /ID# 248783, Osaka, Osaka
  - Japanese Red Cross Osaka Hospi /ID# 248784, Osaka, Osaka
  - Daini Osaka Police Hospital /ID# 240560, Osaka, Osaka
  - Osaka Metropolitan University Hospital /ID# 253203, Osaka, Osaka
  - Nippon Life Saiseikai Public Interest Foundation Nippon Life Hospital /ID# 243783, Osaka, Osaka
  - Kindai University Hospital /ID# 250851, Osakasayama-shi, Osaka
  - Osaka Medical and Pharmaceutical University Hospital /ID# 249440, Takatsuki-shi, Osaka
  - Yao Tokushukai General Hospital /ID# 247884, Yao, Osaka
  - Hara Hospital /ID# 244846, 泉大津市, Osaka
  - Saga Medical Center Koseikan /ID# 245816, Saga, Saga-ken
  - Ageo Central General Hospital /ID# 254515, Ageo-shi, Saitama
  - TMG Asaka Medical Center /ID# 238761, Asaka-shi, Saitama
  - Kamifukuoka General Hospital /ID# 247890, Fujimino, Saitama
  - Shinkuki General Hospital /ID# 254516, Kuki-shi, Saitama
  - Saitama Citizens Medical Center /ID# 252573, Saitama-shi, Saitama
  - NHO Saitama National Hospital /ID# 245061, Wako-shi, Saitama
  - Omi Medical Center /ID# 258233, Kusatsu-shi, Shiga
  - Saiseikai Shiga Hospital /ID# 239381, Rittō, Shiga
  - National Hospital Organization Hamada Medical Center /ID# 250858, Hamada, Shimane
  - Shimane University Hospital /ID# 255194, Izumo-shi, Shimane
  - Shimane Prefectural Central Ho /ID# 247895, Izumo-shi, Shimane
  - Masuda Red Cross Hospital /ID# 248780, Masuda-shi, Shimane
  - Shizuoka Saiseikai Genaral Hospital /ID# 239722, Shizuoka, Shizuoka
  - Duplicate_Dokkyo Medical University Hospital /ID# 246764, Shimotsuga-gun, Tochigi
  - Ishibashi General Hospital /ID# 243762, Shimotsuke, Tochigi
  - Tochigi Cancer Center /ID# 249445, Utsunomiya, Tochigi
  - Anan Medical Center /ID# 243781, Anan-shi, Tokushima
  - Tokushima Prefecture Naruto Hospital /ID# 239095, Naruto-shi, Tokushima
  - Tokushima University Hospital /ID# 252572, Tokushima, Tokushima
  - Juntendo University Hospital /ID# 239096, Bunkyo-ku, Tokyo
  - Tokyo Medical And Dental University Hospital /ID# 242178, Bunkyo-ku, Tokyo
  - St.Luke's International Hospital /ID# 248787, Chuo-ku, Tokyo
  - Medical Plaza Edogawa /ID# 244220, Edogawa Ward, Tokyo
  - Edogawa Hospital /ID# 239352, Edogawa-ku, Tokyo
  - Tama Medical Center /ID# 247954, Fuchū, Tokyo
  - Tokyo Metropolitan Children's Medical Center /ID# 252189, Fuchū, Tokyo
  - Fussa Hospital /ID# 240570, Fussa, Tokyo
  - Tama-Hokubu Medical Center /ID# 245879, Higashimurayama-shi, Tokyo
  - Tokyo Metropolitan Geriatric /ID# 249448, Itabashi-ku, Tokyo
  - Duplicate_Teikyo University Hospital /ID# 247896, Itabashi-ku, Tokyo
  - Meirikai Chuo General Hospital /ID# 238751, Kita-ku, Tokyo
  - Showa General Hospital /ID# 258235, Kodaira, Tokyo
  - Duplicate_The Cancer Institute Hospital Of JFCR /ID# 244216, Koto-ku, Tokyo
  - Mishuku Hospital /ID# 239378, Meguro-ku, Tokyo
  - Kosei Chuo General Hospital /ID# 251011, Meguro-ku, Tokyo
  - Toranomon Hospital /ID# 251010, Minato-ku, Tokyo
  - Japanese Red Cross Musashino Hospital /ID# 246765, Musashino-shi, Tokyo
  - Juntendo Univ Nerima Hospital /ID# 250292, Nerima-ku, Tokyo
  - P_Ome Municipal General Hospital /ID# 248778, Ōme, Tokyo
  - Metropolitan Research and Treatment Center for Blood Disorders /ID# 231384, Setagaya Ward, Tokyo
  - National Center for Child Health and Development /ID# 243778, Setagaya-ku, Tokyo
  - Japanese Red Cross Medical Center /ID# 239385, Shibuya-ku, Tokyo
  - NTT Medical Center Tokyo /ID# 240566, Shinagawa-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 252571, Shinjuku-ku, Tokyo
  - Center hospital of the National Center for Global Health and Medicine /ID# 256189, Shinjuku-ku, Tokyo
  - Kawakita General Hospital /ID# 257009, Suginami-ku, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital /ID# 241912, Sumida-ku, Tokyo
  - The Fraternity Memorial Hospital /ID# 251685, Sumida-ku, Tokyo
  - Eiju General Hospital /ID# 243763, Taitō City, Tokyo
  - Toshima Hospital /ID# 240878, 板橋区, Tokyo
  - Tottori Prefectural Central Ho /ID# 245877, Tottori-shi, Tottori
  - Yonago Medical Center /ID# 240572, Yonago-shi, Tottori
  - Tottori University Hospital /ID# 244215, Yonago-shi, Tottori
  - Kurobe City Hospital /ID# 254493, Kurobe-shi, Toyama
  - Kainan Medical Center /ID# 240825, Kainan, Wakayama
  - Naga municipal Hospital /ID# 250259, Kinokawa, Wakayama
  - Social Insurance Kinan Hosp /ID# 251684, Tanabe-shi, Wakayama
  - Wakayama Rosai Hospital /ID# 250293, Wakayama, Wakayama
  - Okitama Public General Hospital /ID# 242710, Higashiokitama-gun, Yamagata
  - Yamagata University Hospital /ID# 246763, Yamagata, Yamagata
  - NHO Iwakuni Clinical Center /ID# 242170, Iwakuni-shi, Yamaguchi
  - Tokuyama Central Hospital /ID# 242380, Shunan-shi, Yamaguchi
  - Yamaguchi University Hospital /ID# 245060, Ube-shi, Yamaguchi
  - Ogori Daiichi General Hospital /ID# 246761, Yamaguchi, Yamaguchi
  - University of Yamanashi Hospital /ID# 246006, Chuo-shi, Yamanashi
  - Inoue Memorial Hospital /ID# 239351, Chiba
  - National Hospital Organization Chiba Medical Center /ID# 266755, Chiba
  - Fujisawa City Hospital /ID# 239375, Fujisawa-shi
  - Harasanshin Hospital /ID# 240881, Fukuoka
  - Hachinohe Red Cross Hospital /ID# 250850, Hachinohe-shi
  - Tokai University Hachioji Hospital /ID# 266804, Hachiōji
  - Higashihiroshima Medical Center /ID# 250849, Higashihiroshima-shi
  - Hiroshima Prefecture Hospital /ID# 252215, Hiroshima
  - Ikeda City Hospital /ID# 266802, Ikeda
  - Kawaguchi Municipal Medical Center /ID# 246080, Kawaguchi-shi
  - Kitakyusyu General Hospital /ID# 244212, Kitakyushu-shi
  - Kyorin University - Mitaka Campus /ID# 243777, Mitaka
  - Nankai Medical Center /ID# 241914, Saiki-shi
  - Saitama City Hospital /ID# 240567, Saitama
  - Nihonkai General Hospital /ID# 242024, Sakata-shi
  - Tachikawa Hospital /ID# 245878, Tachikawa
  - Takatsuki Red Cross Hospital /ID# 266756, Takatsuki
  - Toshiba General Hospital /ID# 250294, Tokyo
  - Toyama Hospital /ID# 243779, Toyama
  - Shonai Hospital /ID# 254514, Yamagata

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Clinical Study Report Synopsis — https://www.abbvieclinicaltrials.com/study/?id=P20-408#additional-resources-section